CLINICAL TRIAL: NCT02850887
Title: Patient Positioning and Airway Management During Endoscopic Retrograde Cholangiopancreatography ERCP and the Effect on Airway Complications and Procedure Outcomes in Patients With Risks for Anesthesia Adverse Events
Brief Title: Patient Positioning and Airway Management During ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201605151
Record Dates: First submitted 2016-07-21; First posted 2016-08-01 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Airway Management
MeSH Terms: interventions — Deep Sedation; Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- general endotracheal anesthesia (Active Comparator): an inhalation anesthetic (substance that blocks pain) technique in which anesthetic and respiratory gases pass through a tube placed in the trachea (throat) via the mouth or nose
  Interventions: Other: general endotracheal anesthesia
- deep sedation without endotracheal intubation (Active Comparator): local anesthesia together with sedation (drug that produces sleep) and analgesia (drug that treats pain) only.
  Interventions: Other: deep sedation without endotracheal intubation

INTERVENTIONS:
Other: general endotracheal anesthesia — sedation with the use of endotracheal intubation
  Arms: general endotracheal anesthesia
Other: deep sedation without endotracheal intubation — deep sedation without endotracheal airway management.
  Other Names: monitored anesthesia care (MAC)
  Arms: deep sedation without endotracheal intubation

SUMMARY:
The aim of this study is to determine the effect of airway management (a set of medical procedures performed to prevent airway blockage and thus ensure an open path between a patient's lungs and the atmosphere) during endoscopic retrograde cholangiopancreatography [(ERCP), a procedure commonly used to treat conditions of the bile ducts and pancreas] and the effect on airway complications (problems), time to biliary cannulation (access into bile duct) and total procedure duration (length of time). Two methods are being compared and studied: 1) general endotracheal anesthesia: an inhalation anesthetic (substance that blocks pain) technique in which anesthetic and respiratory gases pass through a tube placed in the trachea (throat) via the mouth or nose vs 2) deep sedation without endotracheal intubation: local anesthesia together with sedation (drug that produces sleep) and analgesia (drug that treats pain) only.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing ERCP without preceding endoscopic ultrasound (EUS)
2. At least one of the following risk factors for adverse events during sedation:

   1. STOP-BANG score of 3 or higher
   2. Abdominal ascites on either physical exam or imaging within the last 14 days
   3. BMI greater than or equal to 35
   4. Chronic lung disease
   5. ASA class 4
   6. Mallampati Class 4 airway (only hard palate visible)
   7. Concurrent moderate to heavy alcohol use (≥4 drinks/day for men and ≥3 drinks/day for women)

Exclusion Criteria:

1. EUS preceding the ERCP
2. Emergent indication for ERCP (eg cholangitis with septic shock)
3. Presence of a tracheostomy
4. Unstable airway
5. Gastric outlet obstruction
6. Altered foregut anatomy (eg Roux-en-Y gastric bypass, Billroth II)
7. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of sedation related adverse events or the need for airway maneuvers | approximately one year

SECONDARY OUTCOMES:
Procedure duration | intraoperative
Time to cannulation of intended duct system | during the procedure
Technical success of ERCP | approximately one year
Immediate ERCP adverse events | Adverse events within 24 hours of ERCP
Delayed adverse events | Adverse events occurring within 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith ZL, Mullady DK, Lang GD, Das KK, Hovis RM, Patel RS, Hollander TG, Elsner J, Ifune C, Kushnir VM. A randomized controlled trial evaluating general endotracheal anesthesia versus monitored anesthesia care and the incidence of sedation-related adverse events during ERCP in high-risk patients. Gastrointest Endosc. 2019 Apr;89(4):855-862. doi: 10.1016/j.gie.2018.09.001. Epub 2018 Sep 11. PMID 30217726